CLINICAL TRIAL: NCT05188820
Title: Comparison of IntraArticular Platelet-Rich-Plasma to Corticosteroid Injections for Patients With Zygapophyseal Joint (Z-Joint) Low Back Pain Confirmed by Dual Intra-Articular Local Anesthetic Injections: A Triple Blinded Randomized Controlled Trial
Brief Title: Comparison of IntraArticular Platelet-Rich-Plasma to Corticosteroid Injections for Patients With Zygapophyseal Joint (Z-Joint) Low Back Pain Confirmed by Dual Intra-Articular Local Anesthetic Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Spine Intervention Society (Unknown); Association Québécoise Médecine Sportive et Exercice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21.246
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Platelet Rich Plasma; Zygapophyseal Joint Arthritis
Keywords: low back pain; platelet rich plasma; Zygapophyseal Joint Arthritis
MeSH Terms: conditions — Low Back Pain | interventions — Cortisone

STUDY DESIGN:
Intervention Model Description: Study Design: Triple-blinded randomized controlled trial Patient Sample: Fifty participants with radiological signs of osteoarthritis and Z-Joint LBP confirmed by dual intra-articular local anesthetic injections will be recruited and randomized in two groups: CS and LP-PRP injection groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid group (Active Comparator): Patients will receive intra-articular z-joint injection of cortisone
  Interventions: Procedure: Cortisone injection
- PRP group (Experimental): Patients will receive intra-articular z-joint injection of PRP
  Interventions: Procedure: PRP - platelet rich plasma injection

INTERVENTIONS:
Procedure: PRP - platelet rich plasma injection — Facet block using PRP
  Arms: PRP group
Procedure: Cortisone injection — Facet block using cortisone
  Arms: Corticosteroid group

SUMMARY:
Comparison of IntraArticular Platelet-Rich-Plasma to Corticosteroid Injections for Patients with Zygapophyseal Joint (Z-Joint) Low Back Pain Confirmed by Dual Intra-Articular Local Anesthetic Injections: A Triple Blinded Randomized Controlled Trial.

DETAILED DESCRIPTION:
Abstract/Project Summary Background: Zygapophyseal joint (Z-joint) pain represents up to 40% of lower back pain (LBP), a very common and disabling health issue. There are currently two treatment options for patients with Z-joint LBP unresponsive to conservative treatment: corticosteroid (CS) injections and radiofrequency ablation. CS injection is a shorter, less invasive and readily available procedure. Despite its accepted use, it has not shown its efficacy over placebo.

The use of platelet-rich plasma (PRP) has been investigated for LBP treatment. PRP injection has the same advantages as CS and recent studies suggest that PRP injections are more effective than cortisone from two to six months post treatment. However, no blinded controlled trials have compared these two treatments, and no data is available on the efficacy of PRP after six months for LBP treatment.

Purpose: The purpose of this study is to compare the effect of intra-articular leucocyte poor (LP) PRP to CS injections on pain, function and quality-of-life at 1, 3, 6, 9 and 12month post treatment. The two main outcomes will be the ODI score improvement and the proportion of participants who needs a second injection in each group at one year post treatment.

Study Design: Triple-blinded randomized controlled trial Patient Sample: Fifty participants with radiological signs of osteoarthritis and Z-Joint LBP confirmed by dual intra-articular local anesthetic injections will be recruited and randomized in two groups: CS and LP-PRP injection groups.

Method: Participants will be assessed in person, by mail or by phone at baseline and at 1, 3, 6, 9 and 12-months post-treatment by a blinded evaluator. Pain will be assessed by a visual analogue scale (VAS) when bending over, function by the Oswestry Low Back Disability Index (ODI), quality of life by the SF36 questionnaire and satisfaction by the Modified McNabb Scale.

ELIGIBILITY:
Inclusion Criteria:

* - 40 years old or more; given the low prevalence of facet pain in younger adults
* LBP present for more than six months, with an axial predominance
* Persistent LBP after three months of non-interventional treatment
* Pretreatment ODI score of at least 30/100 (moderate disability associated with LBP)
* Pretreatment LBP VAS of at least 4/10
* 80% LBP reduction 30 minutes after 2 intra-articular diagnostic blocs with Xylocaine and Marcaine
* Radiological signs of facet joint degeneration (on X-rays, CT Scan or MRI)
* Absence of neurological deficit
* Sufficient knowledge of French or English to complete the questionnaires

Exclusion Criteria:

* - Less than 40 years old
* Failure to achieve intra-articular diagnostic block
* Intra-articular injection of CS 3 months or less before recruitment
* Oral corticosteroid use in the last two weeks
* Inflammatory disease
* Systemic infection
* Infection at injection site
* Vertebral fracture
* Spine tumour
* Surgical intervention at injection site prior to the study or planned
* Cognitive disorder that impairs the ability to answer the questionnaires
* Pregnancy
* Breastfeeding
* Coagulopathy affecting platelets
* Drug affecting platelets that cannot be stopped (except acetylsalicylic acid)
* Intolerance or allergies to local anesthetics, contrast agent, CS, and blood products

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale (VAS) | 0, 3, 9, 12 months
  visual analogue scale of pain scale from 0-10 (higher is worse)

SECONDARY OUTCOMES:
Change in Oswestry low back disability index | 0, 3, 9, 12 months
  function due to back pain scale 0-100 (higher is worse)
Change in Short Form 36 scale | 0, 3, 9, 12 months
  quality of life scale score from 0-100 (higher is better)
Change in Modified McNabb scale | 0, 3, 9, 12 months
  satisfaction score 1-5 (higher is better)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hopsitalier Université de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cauchon AM, Mares C, Fan XY, Bois MC, Hagemeister N, Noiseux N, Roy A. Comparing the efficacy of intra-articular injection of Platelet Rich Plasma (PRP) with corticosteroids (CS) in patients with chronic zygapophyseal joint low back pain confirmed by double intra-articular diagnostic blocks: A triple-blinded randomized multicentric controlled trial with a 6-month follow-up. Interv Pain Med. 2024 Dec 3;3(4):100525. doi: 10.1016/j.inpm.2024.100525. eCollection 2024 Dec. PMID 39717452